CLINICAL TRIAL: NCT04905433
Title: The Need for Breathing Retraining: the Elephant in the Cardiac Rehabilitation Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecturer of physical therapy for cardiopulmonary disorders, Faculty of Physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT and CR
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; inspiratory muscle training; cardiac rehabilitation
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation with breathing retraining (Experimental): A cardiac rehabilitation program for 3 days/week (day after day) for 12 weeks(including aerobic, and resisted exercise, with educational sessions, and counseling), with a breathing retraining (using breathing calisthenics, and inspiratory muscle training)
  Interventions: Behavioral: Cardiac rehabilitation with breathing retraining
- cardiac rehabilitation (Active Comparator): A cardiac rehabilitation program for 3 days/week (day after day) for 12 weeks(including aerobic, and resisted exercise, with educational sessions, and counseling) only
  Interventions: Behavioral: Cardiac rehabilitation

INTERVENTIONS:
Behavioral: Cardiac rehabilitation with breathing retraining — A cardiac rehabilitation program for 3 days/week (day after day) for 12 weeks(including aerobic, and resisted exercise, with educational sessions, and counseling), with a breathing retraining (using breathing calisthenics, and inspiratory muscle training)
  Arms: Cardiac rehabilitation with breathing retraining
Behavioral: Cardiac rehabilitation — A cardiac rehabilitation program for 3 days/week (day after day) for 12 weeks(including aerobic, and resisted exercise, with educational sessions, and counseling) only
  Arms: cardiac rehabilitation

SUMMARY:
As an extension of previous work, in this study, a breathing retraining component is added using breathing calisthenics and inspiratory muscle trainer for the classical cardiac rehabilitation (CR), as an appealing option, to implement a comprehensive rehabilitation protocol addressing the different patient-centered outcomes including different cardiovascular, and respiratory complaints; increasing the benefits of classical CR; detecting the impact of adding this on the cardiovascular (CV) outcomes, and discovering the correlation between the CV and respiratory data.

DETAILED DESCRIPTION:
A very large number of studies have demonstrated the positive effect of cardiac rehabilitation (CR) and pulmonary rehabilitation (PR) on morbidity and mortality. Globally, each year millions of patients with different cardiovascular diseases (CVD) and chest diseases are enrolled in these programs. The exact effects may be slightly variable, but generally, both CR and PR aim to improve the patient's condition and improve the overall quality of life utilizing almost the same methods (exercise, and education).

Despite these positive effects, utilization rates of either CR or PR are around 30% in Europe, with much less percentages in the Middle East. The reasons for the low engagement rates are many; with most probably the main reasons are about individuality and reach. Optimized CR programs have to be individually tailored; meeting the individual needs of every single patient in the program. Worse knowing that the chest pain and breathlessness are highly prevalent in general in CVD, and considered -in many cases as the chief complaint, and the classical CR programs are neglecting these complaints; negatively affecting adherence rates and patient-centered outcomes (PCO) which mostly extend much beyond the cardiovascular complaints, to extend to the respiratory, and sleep complaints; questioning the reason why breathing retraining methods are not yet considered as an integral part of the CR programs.

The reason that standard CR programs usually neglect these complaints, and only look for the CV outcomes; is considering the other mentioned complaints as "out-of-context". However, solid evidence is suggesting a strong correlation between respiratory, sleep, and CV outcomes.

It has been previously investigated the impact of the CR on sleep, and there is a prior estimate suggesting that 25% of the participants in the CR programs have already sleep disorders, there is a strong correlation between the sleep and CV outcomes, and almost all of the patients in the CR have respiratory symptoms including dyspnea and functional capacity decline.

Therefore, it was suggested adding a breathing retraining component using breathing calisthenics and inspiratory muscle trainer for the classical CR, as an appealing option, to implement a comprehensive rehabilitation protocol addressing the different PCO including different cardiovascular, and respiratory complaints; increasing the benefits of classical CR; detecting the impact of adding this on the CV outcomes, and discovering the correlation between the CV and respiratory data.

ELIGIBILITY:
Inclusion Criteria:

* . chronic heart failure (≥ 1 year) .Respiratory muscle weakness≤ 70% of their predicted MIP.

  * Ages ranged from 45-65 years old
  * Left ventricle ejection fraction ≤ 40% in NYHA class II and III .In stable condition (No rales on auscultation or tibial edema and with sinus rhythm).
  * On standard cardiac medications (diuretics, angiotensin-converting enzyme (ACE) inhibitors, and glycosides)
  * Not engaged in any regular physical training program for at least one month before the start of the study.

Exclusion Criteria:

* Chronic lung disorders,

  * Anemia
  * Severe hypoxia
  * History of myocardial infarction or pulmonary edema six months before the study
  * Severe uncontrolled hypertension, or uncontrolled diabetes mellitus or autonomic disorders

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
heart rate variability | 12 weeks
  represent autonomic response of the heart (measured through a holter ECG)
functional capacity | 12 weeks
  represents aerobic fitness (VO2 max) (ml/kg/min) measured through cardiopulmonary exercise testing
anaerobic threshold | 12 weeks
  represents lactate threshold (% of VO2 max) measured through cardiopulmonary exercise testing
resting heart rate | 12 weeks
  represents resting condition of the heart (beat/min)
resting systolic blood pressure | 12 weeks
  represents resting condition of the systolic blood pressure (mmhg) measured by sphygmomanometer
resting diastolic blood pressure | 12 weeks
  represents resting condition of the diastolic blood pressure (mmhg) measured by sphygmomanometer

SECONDARY OUTCOMES:
forced vital capacity | 12 weeks
  represents volume of air in a forced expiration after full inspiration (%) measured by pulmonary function testing
rate of perceived exertion | 12 weeks
  represents level of patient exertion on exercise measured by modified Borg scale (1-10), where lower scores means lower levels of exertion, and higher scores means higher levels of exertion.

CONTACTS AND LOCATIONS:
Overall Officials: Hady Atef, PhD, Principal Investigator — Cairo University, Egypt; Donna Fitzimons, Prof, Study Director — Queen's University, Belfast
Locations (1):
- National heart institute, Cairo, AI Qahirah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After approval can be shared
Supporting Information: Study Protocol
Time Frame: after 1 month for12 months
Access Criteria: will upload it to the journal of publication